CLINICAL TRIAL: NCT00403195
Title: Pathophysiological Analysis of Ocular Ischemic Syndrome and the Response to Vascular Surgery
Brief Title: Clinical and Pathophysiological Description of Ocular Ischemic Syndrome
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Kofoed, Principal investigator, Glostrup University Hospital, Copenhagen
Other Study IDs: OIS
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Retinal Degeneration; Diabetic Retinopathy
Keywords: Ocular Ischemic Syndrome
MeSH Terms: conditions — Retinal Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize the disease Ocular Ischemic Syndrome.

DETAILED DESCRIPTION:
The disease Ocular Ischemic Syndrome (OIS) is not a well described entity. It occurs after a long-standing period of extremely low blood supply to the retina caused by atherosclerosis of the carotid arteries. In this study we will analyze why OIS is developed in some patients and not developed in others. The patients with OIS will be thorough examined and will be compared with 1) a control group of healthy people and 2) with control group of patients with diabetic retinopathy. Furthermore the impact of vascular surgery on OIS will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ocular ischemic syndrome

Exclusion Criteria:

* Any other active ocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with the disease ocular ishemic syndrome. Patients will be screened through vascular surgery departments.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larsen, Professor, Study Director
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Kofoed PK, Munch IC, Sander B, Holfort SK, Sillesen H, Jensen LP, Larsen M. Prolonged multifocal electroretinographic implicit times in the ocular ischemic syndrome. Invest Ophthalmol Vis Sci. 2010 Apr;51(4):1806-10. doi: 10.1167/iovs.09-4555. Epub 2009 Nov 20. PMID 19933192